CLINICAL TRIAL: NCT00708630
Title: The Effect of Extended Yellow Fever Vaccine Information on Symptom Reports Following Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Keith J Petrie, Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: KPKF001
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Vaccination
Keywords: yellow fever vaccine; patient information; symptom reports; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Provision of extended symptom side effects information
  Interventions: Behavioral: Extended information on side effects
- 2 (No Intervention): Standard information on side effects

INTERVENTIONS:
Behavioral: Extended information on side effects — More detailed information on possible side effects of vaccine
  Arms: 1

SUMMARY:
This study aims to investigate the effect of providing additional information about possible mild side effects of the yellow fever vaccination on the reporting of physical symptoms. Additionally, the project aims to investigate the relationship between individual characteristics (trait anxiety and perceived sensitivity to medication) and the reporting of physical symptoms, as well as possible interactions between the level of information provided and individual characteristics. We hypothesize that more information about mild symptoms provided to participants will increase the number of reported symptoms after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Receiving yellow fever vaccination
* English speaker
* Aged over 18

Exclusion Criteria:

* No phone for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
symptom report scale | 20 minutes and 1 week post vaccination

SECONDARY OUTCOMES:
patient satisfaction scale | 20 minutes and 1 week post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Keith J Petrie, PhD, Principal Investigator — University of Auckland, New Zealand; Kate E Faasse, BSc, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Worldwise Travellers Health, Auckland, Auckland, New Zealand